CLINICAL TRIAL: NCT00727220
Title: A Prospective Study of the Impact of CSII Therapy in Young Children With Type 1 DM
Brief Title: Prospective Study of the Impact of Insulin Pump Therapy in Young Children With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Linda DiMeglio, MD, MD, Indiana University
Other Study IDs: 0312-13
Record Dates: First submitted 2008-07-30; First posted 2008-08-01 (Estimated); Results first posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; continuous glucose sensor monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Insulin Pump Therapy: Children starting insulin pump therapy
- Insulin Injections: Children remaining on insulin injections.

SUMMARY:
The purpose of the study is to examine glycemic and neuropsychological outcomes in very young children with Type I diabetes who are being started on insulin pumps and to compare their outcomes to children who are not utilizing insulin pumps. We propose to assess 40 children with IDDM under 5 years of age. 10 patients examined will be using multiple daily injections with basal glargine, 10 will be using NPH or Lente and rapid-acting insulin, and 20 will be examined prior to and 12 months after the implementation of insulin pump therapy. These subjects will be recruited and followed because they are currently undergoing treatment for Type 1 diabetes. Children will be recruited based upon the insulin regimen that they and their primary diabetes physician have chosen to utilize clinically. Insulin regimens will not be changed by the study team. Outcome measures will examine: glycemic outcomes (overall control, blood sugar variability), cognitive outcomes, parenting Stress, and changes in diet.

ELIGIBILITY:
Inclusion Criteria:

1. Children with Type I diabetes:
2. Children must be 5 years of age or less at the time of entry into the study.
3. Children must have had a diagnosis of type I diabetes for at least 1 year at time of entry.
4. Children must be receiving two or more insulin injections daily.

Exclusion Criteria:

1. Children will be excluded if they have additional medical problems requiring treatment with agents known to affect blood glucose such as steroids or L-asparaginase.
2. Children must not have any other chronic illness in addition to diabetes.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children diagnosed with type 1 diabetes for at least one year at the time of study. In addition, children must be under the age of 5 years
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 1999-11; Primary Completion 2003-04 (Actual); Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda DeMeglio, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Riley Hospital for Children, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Insulin Pump Therapy | Insulin Injections
Started | 21 | 21
Completed | 20 | 17
Not Completed | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Pump Therapy | Insulin Injections | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21 | 21 | 42
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.8 (0.8) | 3.7 (0.7) | 3.8 (0.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 25
  Male | 10 | 7 | 17
Region of Enrollment [Number; unit: participants]
  United States | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: Change in HgBA1c
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Insulin Pump Therapy | Insulin Injections
Number analyzed (Participants) | 20 | 17
percentage of glycosylated hemoglobin | 8.5 (0.6) | 8.7 (0.7)

ADVERSE EVENTS:
Arm/Group | Insulin Pump Therapy | Insulin Injections
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes